CLINICAL TRIAL: NCT07355140
Title: Comparative Study of Vital Pulp Therapy and Root Canal Treatment in Mature Permanent Teeth With Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Vital Pulp Therapy vs. Root Canal Treatment in Mature Teeth With Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Central de Venezuela (Other)
Responsible Party: Principal Investigator, Juan Norberto Goncalves Pereira, Clinical Professor, Universidad Central de Venezuela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UCVenezuela
Record Dates: First submitted 2026-01-04; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pulpitis - Irreversible; Pulpitis; Pulpotomy; Root Canal Therapy
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled, parallel-group, double-blind clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vital Pulp Therapy Group (VPT Group) (Experimental): A 10 mL blood sample was collected to obtain PRF following Choukroun's protocol. Caries removal was performed non-selectively using sterile carbide burs at high speed with water cooling. After pulp exposure, passive irrigation with 5.25% NaOCl was performed. Inflamed pulp tissue was gradually removed under magnification using a fine-grit diamond bur until vascular, slightly bleeding tissue was observed. Hemostasis was achieved by gentle pressure with a sterile dry cotton pellet; if bleeding persisted, additional tissue removal was performed for up to 15 minutes. In some cases, full pulpotomy was required. PRF was compressed and trimmed to cover the exposed pulp tissue, then sealed with 2-3 mm of EndoSequence BC putty. The cavity was restored with self-curing glass ionomer and definitive composite resin.
  Interventions: Procedure: VPT Group and RCT Group
- Root Canal Treatment Group (RCT Group) (Active Comparator): After caries removal, access cavity preparation was performed, and working length was determined using an electronic apex locator (Root ZX; J Morita, Irvine, CA). Root canals were instrumented with nickel-titanium rotary files (.04 taper) up to three sizes beyond the first file, with resistance. Irrigation was performed with 5.25% NaOCl and 17% EDTA. Obturation was completed using lateral compaction with gutta-percha and AH Plus sealer. The access cavity was sealed with glass ionomer and restored with composite resin.
  Interventions: Procedure: VPT Group and RCT Group

INTERVENTIONS:
Procedure: VPT Group and RCT Group — In the VPT group, partial or complete pulpotomy was performed using PRF, followed by a bioceramic covering and definitive restoration. In the RCT group, root canal treatment was performed, and the coronal access was definitively sealed.

SUMMARY:
This study was designed as a prospective, randomized, controlled clinical trial with parallel groups and double blinding, following the principles of the Declaration of Helsinki for human experimentation and in accordance with CONSORT guidelines. The study protocol was approved by the Bioethics Committee of the Faculty of Dentistry, Central University of Venezuela

Forty-six patients were enrolled and evenly assigned to two groups (VPT group: Vital Pulp Therapy Group; RCT Group: Root canal treatment group); 43 completed the 12-month follow-up (22 in the VPT group and 20 in the RCT group).

Patients were assigned to the experimental group (VPT) or control group (RCT) using a block randomization method (block size = 4). The randomization sequence was kept in sealed envelopes and revealed by a team member not involved in the study.

Clinical Procedures:

Preoperative periapical radiographs were taken using the parallel cone technique for both groups, and bitewing radiographs were additionally obtained for the experimental group. All procedures were performed under local anesthesia with 3% mepivacaine (inferior alveolar nerve block for mandibular teeth and infiltration for maxillary teeth) and rubber dam isolation.

* Experimental Group (VPT): A 10 mL blood sample was collected to obtain PRF following Choukroun's protocol. Caries removal was performed non-selectively using sterile carbide burs at high speed with water cooling. After pulp exposure, passive irrigation with 5.25% NaOCl was performed. Inflamed pulp tissue was gradually removed under magnification using a fine-grit diamond bur until vascular, slightly bleeding tissue was observed. Hemostasis was achieved by gentle pressure with a sterile dry cotton pellet; if bleeding persisted, additional tissue removal was performed for up to 15 minutes. In some cases, full pulpotomy was required. PRF was compressed and trimmed to cover the exposed pulp tissue, then sealed with 2-3 mm of EndoSequence BC putty. The cavity was restored with self-curing glass ionomer and definitive composite resin.

* Control Group (RCT): After caries removal, access cavity preparation was performed, and working length was determined using an electronic apex locator (Root ZX; J Morita, Irvine, CA). Root canals were instrumented with nickel-titanium rotary files (.04 taper) up to three sizes beyond the first file, with resistance. Irrigation was performed with 5.25% NaOCl and 17% EDTA. Obturation was completed using lateral compaction with gutta-percha and AH Plus sealer. The access cavity was sealed with glass ionomer and restored with composite resin.

ELIGIBILITY:
Inclusion Criteria:

* Posterior teeth with closed apices.
* Deep carious lesions radiographically close to the pulp.
* Symptoms of symptomatic irreversible pulpitis (spontaneous and/or sharp pain, localized or referred, provoked and persistent to thermal stimuli).
* Teeth restored with direct restorations.

Exclusion Criteria:

* Subgingival caries or restorations.
* Moderate or severe periodontitis.
* Internal or external resorption.
* Calcification of the pulp chamber or root canals.
* Uncontrolled pulpal bleeding within 15 minutes.

Ages: 26 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Teeth Categorized as Clinical and Radiographic Success | 12 months
  Success is a composite measure defined by the following criteria:
  Clinical Success: Absence of spontaneous pain (excluding the immediate postoperative period), tooth is functional and asymptomatic, with no sensitivity to percussion or palpation, and normal soft tissues.
  Radiographic Success: Absence of periapical pathology, such as new periapical radiolucency or root resorption.
  A case is considered a "Success" only when both clinical and radiographic criteria are met. Results will be reported as the percentage of teeth that meet these success criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Central University of Venezuela, Caracas, DC, Venezuela

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available starting 6 months and up to 1 year following article publication